CLINICAL TRIAL: NCT07402356
Title: Task-evoked Pupillometry in AD, MCI, and Depression-Related Cognitive Impairment
Brief Title: VR Pupillometry in Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Principal Investigator, Victor Spoormaker, Principal Investigator, Max-Planck-Institute of Psychiatry
Other Study IDs: 23-0991
Record Dates: First submitted 2026-01-12; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer s Disease; Major Depressive Disorder (MDD); Mild Cognitive Impairment; Dementia
Keywords: Alzheimer's Disease; Major Depressive Disorder; Mild Cognitive Impairment; Dementia; Pupillometry; Biomarkers; Amyloid beta-Peptides; Tau Proteins
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction; Dementia; Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and CSF; for marker analyses + control/calibration; Optional biobank opt-in (Munich Mental Health Biobank)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Alzheimer's Disease: Participants with complaints of cognitive deficits and a diagnosis of Alzheimer's disease (AD) supported by cerebrospinal fluid (CSF) biomarker profile, where available.
- Mild Cognitive Impairment without Alzheimer's Disease: Participants with complaints of cognitive deficits meeting criteria for mild cognitive impairment without evidence of Alzheimer's disease (CSF biomarkers not consistent with AD).
- Depressive Disorder With Cognitive Impairment: Participants with complaints of cognitive impairment and no evidence of Alzheimer's pathology; deficits most consistent with depressive disorder.
- Healthy Controls: Age-matched healthy volunteers.

SUMMARY:
With disease-modifying therapies emerging for dementia and related conditions, identifying cognitive decline as early as possible is increasingly important. This prospective, single-center, repeated-measures study evaluates whether VR-based eye-tracking pupillometry can provide a practical, non-invasive biomarker of cognitive impairment and its progression over time. Pupil responses are linked to brain arousal systems relevant to cognitive dysfunction, including the locus coeruleus, which is affected early in Alzheimer's disease. Adults aged 18-80 years will be assigned to one of four cohorts (n=35 per cohort): i) Alzheimer's disease (supported by CSF biomarkers), ii) mild cognitive impairment (MCI) without Alzheimer's Disease, iii) depressive disorder with cognitive impairment, iv) healthy controls. Participants will undergo initial assessments at baseline and follow-up visit after 3 and 6 months. At each visit, pupil responses and behavioral metrics are recorded during a pupillary light reflex paradigm, a resting-state fixation block, a working-memory task (N-back), and a reward task. Pupillometric and behavioral metrics will be compared across cohorts and related to routine neuropsychological measures (MoCA, CERAD) and available clinical biomarkers (CSF markers; blood biomarkers). The primary objective is to determine whether task-evoked pupil response profiles sensitively quantify cognitive impairment, differ between cohorts, and track change over time. The long-term goal is to validate an easy-to-use, outpatient-compatible assessment to support objective characterization and monitoring of cognitive disorders.

DETAILED DESCRIPTION:
Cognitive performance typically declines with age and is usually accompanied by attention and memory deficits. While such changes can be consistent with normal ageing, they may also reflect affective disorders or early stages of neurodegenerative diseases (e.g. Alzheimer's Disease; AD). In clinical practice, neurocognitive tests are commonly used to distinguish age-appropriate change from pathological decline. As these tests quantify behavioral performance, they are better at detecting cognitive decline, once measurable deficits are manifested. However, they have limited sensitivity to subtle changes that can precede overt clinical symptoms by several years. We therefore propose a simple diagnostic approach based on pupil dilation measurements that may support earlier detection and longitudinal monitoring, potentially enabling earlier interventions.

Pupillometry provides a noninvasive index of pupil dynamics linked to arousal systems relevant to cognition, including the locus coeruleus-noradrenergic (LC-NA) system. LC-NA activity is coupled to pupil dilation via autonomic pathways, and this coupling has been demonstrated across animal and human studies. Given its widespread projections, the LC-NA system is implicated in psychiatric and neurological conditions through roles in arousal regulation, stress responsivity, attention, and memory. Pupillometry in Alzheimer's disease has often been examined using pupillary light reflex paradigms. However, simple light-flash measures may be less informative in early-stage impairment because pupil responses vary with cognitive state and task demands and do not provide a uniform, task-independent readout of LC-linked function. Accordingly, analyzing pupil responses during and immediately following cognitive tasks may be better suited to capturing subtle dysfunction relevant to prodromal processes, with light-reflex alterations potentially becoming more apparent once impairment is established. In prior work, we observed pupil diameter increased with working-memory load during an N-back task. Most participants showed the expected increase in pupil dilation with task difficulty, whereas a subset exhibited pronounced atypical pupil responses despite only slight differences on standard neurocognitive measures. Building on these principles, this study uses a VR-based assessment to examine adults presenting with early, non-specific cognitive complaints. By systematically recording pupil dynamics during and following cognitive paradigms, we aim to obtain readouts of LC-NA system function that may support differential diagnosis among conditions with overlapping clinical presentations (e.g. depression-related cognitive impairment vs. early dementia).

At each visit, participants are fitted with a VR headset by trained study personnel and complete VR-based assessments with concurrent eye tracking and behavioral performance recording. Assessments are conducted at baseline (T0) and repeated after 3 months (T1) and 6 months (T2). At each visit, pupil responses and task performance are recorded during a pupillary light reflex paradigm, a resting-state fixation block, a working-memory task (N-back), and a reward task. Participants also complete routine neuropsychological testing, including the Montreal Cognitive Assessment (MoCA) and the CERAD battery comprising semantic fluency, Boston Naming Test, Mini-Mental State Examination (MMSE), word list learning, word list delayed recall, word list recognition, figure copying, figure delayed recall, phonemic fluency, and Trail Making Test. Additional assessments include the Bayer Activities of Daily Living scale (Bayer-ADL) and the Geriatric Depression Scale (GDS), as well as questionnaires assessing subjective cognitive impairment (FLei) and childhood adversity (CTQ). Sociodemographic data are recorded, including age, sex, education (years of schooling), and occupation. Blood is collected for routine laboratory measures and blood-based biomarker analyses (including phosphorylated tau 217), and clinical data from routine care are linked where available. In some cases, cerebrospinal fluid biomarkers from routine clinical evaluation are available and linked, including AD pathology markers (amyloid-β and tau measures).

Pupillometric and behavioral measures will be compared across cohorts and evaluated longitudinally across follow-up visits. Measures will also be related to routine neuropsychological assessment, as well as available clinical biomarkers (CSF amyloid-β and tau measures blood-based biomarkers and anatomical neuroimaging sequences). Our prior observations suggest that pupil dilation scales with cognitive load and that task-evoked pupil responses can differ, even when standard neurocognitive measures show only subtle differences. We hypothesize that task-evoked pupil response patterns will differ between cohorts and may be sensitive to change over time.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age 18-80 years.
3. Ability to read and understand German.
4. For patient cohorts: suspected or confirmed diagnosis of AD/MCI/depressive disorder with cognitive impairment according to clinical assessment and routine documentation.

Exclusion Criteria:

1. Acute suicidality (e.g. BDI suicidality item > 1).
2. Change of psychotropic medication within the last 4 weeks.
3. Lifetime psychotic disorder (ICD-10 F20-29).
4. Lack of capacity to consent.
5. Lifetime bipolar disorder (ICD-10 F31).
6. Acute substance abuse or harmful use of alcohol or other psychoactive substances.
7. Parkinson's syndrome (ICD-10 G20).
8. Multiple sclerosis (ICD-10 G35).
9. Stroke within the last 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-80 years will be recruited at the Max Planck Institute of Psychiatry (Munich, Germany) from inpatient wards and outpatient clinics. Patients have a suspected or confirmed clinical diagnosis of Alzheimer's disease, mild cognitive impairment, or depressive disorder with cognitive impairment. Routine clinical measures (neuropsychological testing and, CSF biomarkers, blood biomarkers, imaging) will be linked to study pupillometry outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Task-evoked pupil dilation during N-Back | Baseline
  Pupil response metrics (mean relative pupil diameter in each condition) recorded with VR eye tracking during the N-back task for each condition (fixation, 0-back, 1-back, 2-back, 3-back).

SECONDARY OUTCOMES:
Resting-state pupil dynamics | Baseline, 3 months, 6 months.
  Mean and variability of pupil diameter during resting fixation.
Reward-task pupil response | Baseline, 3 months, 6 months.
  Pupil response metrics (mean relative pupil diameter in each condition) recorded with VR eye tracking during each condition (reward, control).
N-back behavioral performance | Baseline, 3 months, 6 months.
  Behavioral performance during the VR N-back task, quantified as accuracy and reaction time for each load condition (0-, 1-, 2-back).
Montreal Cognitive Assessment (MoCA) | Baseline, 3 months, 6 months.
  Global cognitive screening tool used to quantify overall cognitive impairment.
CERAD cognitive battery | Baseline, 6 months.
  CERAD subtests: semantic fluency (animals), Boston Naming Test, word list learning (immediate recall across trials), word list delayed recall, word list recognition, figure copying, figure delayed recall, phonemic fluency (S-words), and Trail Making Test.
Bayer Activities of Daily Living | Baseline, 6 months.
  Functional status measured using the Bayer-ADL total score, reflecting deficits in the performance of everyday activities.
Geriatric Depression Scale | Baseline, 6 months.
  Depressive symptom severity measured using the GDS total score.
Subjective cognitive impairment | Baseline, 6 months.
  Self-reported subjective cognitive impairment assessed using the Mental Capacity Questionnaire (FLei) total score
Childhood Trauma Questionnaire | Baseline.
  Retrospective recall-based measures administered to adults. Used to determine experiences of childhood trauma.
Blood-based biomarkers | Baseline, 6 months.
  Blood biomarker concentrations assessed from collected blood samples, including phosphorylated tau 217 (p-tau217) and Aβ1-42/Aβ1-40 ratio.
CSF Alzheimer's disease pathology markers | Baseline.
  CSF biomarkers from routine clinical evaluation where available, including Aβ1-42, Aβ1-40, Aβ1-42/Aβ1-40 ratio, total tau, and phosphorylated tau.
Task-evoked pupil dilation during N-Back. | 3 months, 6 months.
  Pupil response metrics (mean relative pupil diameter in each condition; load-dependent slope across conditions) recorded with VR eye tracking during the N-back task for each condition (fixation, 0-back, 1-back, 2-back, 3-back).

OTHER OUTCOMES:
Between-group differences in N-back pupil metrics | Baseline, 3 months, 6 months.
  Comparison of the primary N-back pupil load metric across the four cohorts (Alzheimer's disease, mild cognitive impairment, depressive disorder with cognitive impairment, healthy controls).
Association between task-evoked pupil responses and cognitive test performance | Baseline, 6 months.
  Association between the N-back pupil metrics and cognitive performance measures (MoCA total score; CERAD).
Association between task-evoked pupil responses and AD pathology markers | Baseline through 6 months, using biomarker time points available
  Association between the N-back pupil metrics and available biomarkers of AD pathology (CSF and blood-based biomarkers).
Change from baseline in N-back pupil metrics | Baseline, 3 months, 6 months.
  Within-participant change from baseline in the prespecified N-back pupil load metric

CONTACTS AND LOCATIONS:
Overall Officials: Victor I. Spoormaker, PhD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy PR, O'Connell RG, O'Sullivan M, Robertson IH, Balsters JH. Pupil diameter covaries with BOLD activity in human locus coeruleus. Hum Brain Mapp. 2014 Aug;35(8):4140-54. doi: 10.1002/hbm.22466. Epub 2014 Feb 7. PMID 24510607
- [Background] Megemont M, McBurney-Lin J, Yang H. Pupil diameter is not an accurate real-time readout of locus coeruleus activity. Elife. 2022 Feb 2;11:e70510. doi: 10.7554/eLife.70510. PMID 35107419
- [Background] Fietz J, Pohlchen D; BeCOME Working Group; Bruckl TM, Brem AK, Padberg F, Czisch M, Samann PG, Spoormaker VI. Data-Driven Pupil Response Profiles as Transdiagnostic Readouts for the Detection of Neurocognitive Functioning in Affective and Anxiety Disorders. Biol Psychiatry Cogn Neurosci Neuroimaging. 2024 Jun;9(6):580-587. doi: 10.1016/j.bpsc.2023.06.005. Epub 2023 Jun 20. PMID 37348604
- [Background] Fietz J, Pohlchen D, Binder FP; BeCOME Working Group; Czisch M, Samann PG, Spoormaker VI. Pupillometry tracks cognitive load and salience network activity in a working memory functional magnetic resonance imaging task. Hum Brain Mapp. 2022 Feb 1;43(2):665-680. doi: 10.1002/hbm.25678. Epub 2021 Oct 8. PMID 34622518
- [Background] Aston-Jones G, Cohen JD. An integrative theory of locus coeruleus-norepinephrine function: adaptive gain and optimal performance. Annu Rev Neurosci. 2005;28:403-50. doi: 10.1146/annurev.neuro.28.061604.135709. PMID 16022602